CLINICAL TRIAL: NCT00347646
Title: An Open Label Sequential Dose Response Observational Study of Intravitreally Administered Plasmin for the Creation of a Posterior Vitreous Detachment (PVD)
Brief Title: A Study to Evaluate Plasmin for the Creation of a Posterior Vitreous Detachment (PVD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 484
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Vitreoretinal Traction Syndrome
MeSH Terms: interventions — Fibrinolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasmin (Experimental): Human-derived plasmin reconstituted with sterile sodium chloride for intravitreal injection.
  Interventions: Drug: Plasmin

INTERVENTIONS:
Drug: Plasmin — 27 mg of human-derived plasmin to be reconstituted with of 0.9% Sterile Sodium Chloride for a single intravitreal injection

SUMMARY:
Plasmin is expected to create a posterior vitreous detachment (PVD) when injected directly into the eye. The pharmacological creation of a PVD may be beneficial in helping to treat a variety of conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are in need of a vitrectomy.

Exclusion Criteria:

* A PVD in the study eye as assessed by the investigator using ophthalmic and alternative examination techniques.
* A history of vitrectomy in the study eye.
* A media opacity that precludes quality examination of the vitreous and fundus in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Presence of a Posterior Vitreous Detachment (PVD) | 14 days
  Presence of posterior vitreous detachment evaluated durning virectomy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States